CLINICAL TRIAL: NCT05957952
Title: The Effects of Dynamic Taping With Exercise on Neuromuscular Control
Brief Title: The Effects of Dynamic Taping With Exercise on Neuromuscular Control in Individuals With Subacromial Impingement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112007AF
Record Dates: First submitted 2023-07-02; First posted 2023-07-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder Impingement Syndrome; Transcranial magnetic stimulation; Dynamic tape; Corticospinal system; Scapular control exercise; Kinematics; Muscle activation
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Sham Comparator): Motor control exercise
  Interventions: Procedure: Motor control exercise
- Dynamic taping with exercise group (Experimental): Motor control exercise combined with dynamic taping
  Interventions: Procedure: Motor control exercise with dynamic taping

INTERVENTIONS:
Procedure: Motor control exercise with dynamic taping — Subjects will learn how to control their scapula during motor control exercise with application of dynamic tape
  Arms: Dynamic taping with exercise group
Procedure: Motor control exercise — Subjects will learn how to control their scapula during motor control exercise without taping
  Arms: Exercise group

SUMMARY:
Background: Subacromial Impingement Syndrome (SIS) is the commonest disorder of the shoulder, accounting for 44%-65% of all complaints of shoulder pain. Previous studies have found kinematic changes and alterations in muscle activation amplitude or timing. Recent studies also show the different organization of the corticospinal system in patients with SIS and alterations in central motor representation in individuals with rotator cuff tendinopathy. To restore kinematic changes and muscle activation in patients with SIS, treatments of patients with SIS commonly include motor control exercise and taping. However, there are different types of taping with different properties and purposes resulting in inconsistent outcomes. Recently, a new taping technique, Dynamic tape whose properties are between the most common taping Kinesio tape and rigid tape may solve the questions above. But the evidence of the effect of Dynamic tape and the additional effect of Dynamic tape with motor control exercises are still not well understood. Purpose: The purpose of this study is to investigate the additional effects of Dynamic taping with motor control exercise compared to motor control exercise alone on kinematic, muscle activity, corticospinal excitability, pain and function in people with subacromial Impingement Syndrome.

Methods: This is a randomized control trial. Fifty individuals with SIS will be randomly assigned into either an exercise group or dynamic tape with exercise group. Both groups will receive 5 sessions of treatment in 2 weeks, with 30 minutes per sessions. Outcomes will be measured at baseline, after the first intervention and following 2-week intervention. Primary outcome measures will include scapular kinematics, scapular muscle activation and corticospinal system. Secondary outcome measures included shoulder pain by a numeric pain rating scale and shoulder function by the disability of the arm, shoulder & hand scale (DASH). Data analysis: two-way and three-way mixed ANOVA will used to compare the intervention effect of two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain located on the front or outer side.
2. The participants were only included if they were aged between 20-40 years.
3. Total participation time in shoulder exercises per week is greater than or equal to 4 hours.
4. Presence of scapular movement dysfunction.
5. Presence of shoulder impingement symptoms, with at least 3 positive results in the following 6 tests:

   * Painful arc test
   * Neer's impingement test
   * Hawkins-Kennedy impingement test
   * Empty can test
   * Resisted external rotation test
   * Tenderness of the rotator cuff tendons

Exclusion Criteria

1. Received shoulder exercise therapy in the past three months.
2. Arm elevation angle less than 120 degrees
3. Have a history of dislocation, fracture, or surgery of upper extremity
4. A history of direct contact injury to the neck or upper extremities within the past 12 months
5. A concussion within the past 12 months or a history of three or more concussions
6. Brain injury and neurological impairment
7. History of frequent headache or dizziness
8. Contraindications to the use of transcranial magnetic stimulation, assessed with a safety screening questionnaire, including pregnancy, history of seizure, epilepsy and syncope, having cochlear implant, having medal implant and taking anti-depressant medication.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological measures - Active motor threshold | Change from baseline AMT at the completion of the first 30-minute intervention
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Neurophysiological measures - Active motor threshold | Change from baseline AMT at the completion of 5-session intervention, an average of 2 weeks
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Neurophysiological measures - Motor evoked potential | Change from baseline MEP at the completion of the first 30-minute intervention
  Motor evoked potential (MEP) will be described with millivolt (mV).
Neurophysiological measures - Motor evoked potential | Change from baseline MEP at the completion of 5-session intervention, an average of 2 weeks
  Motor evoked potential (MEP) will be described with millivolt (mV).
Neurophysiological measures - Cortical silent period | Change from baseline CSP at the completion of the first 30-minute intervention
  Cortical silent period (CSP) will be measured with millisecond (ms).
Neurophysiological measures - Cortical silent period | Change from baseline CSP at the completion of 5-session intervention, an average of 2 weeks
  Cortical silent period (CSP) will be measured with millisecond (ms).
Neurophysiological measures - Short interval cortical inhibition | Change from baseline SICI at the completion of the first 30-minute intervention
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Neurophysiological measures - Short interval cortical inhibition | Change from baseline SICI at the completion of 5-session intervention, an average of 2 weeks
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Neurophysiological measures - Short interval cortical facilitation | Change from baseline SICF at the completion of the first 30-minute intervention
  Short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms
Neurophysiological measures - Short interval cortical facilitation | Change from baseline SICF at the completion of 5-session intervention, an average of 2 weeks
  Short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms

SECONDARY OUTCOMES:
Scapular kinematics | Change from baseline scapular kinematics at the completion of the first 30-minute intervention
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plan elevation at 30°, 60°, 90°, and 120°, will be calculated and will be described with degree (°).
Scapular kinematics | Change from baseline scapular kinematics at the completion of 5-session intervention, an average of 2 weeks
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plan elevation at 30°, 60°, 90°, and 120°, will be calculated and will be described with degree (°).
Scapular muscles activation | Change from baseline scapular muscles activation at the completion of the first 30-minute intervention
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°
Scapular muscles activation | Change from baseline scapular muscles activation at the completion of 5-session intervention, an average of 2 weeks
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°
Shoulder function | Change from baseline DASH questionnaire at the completion of 5-session intervention, an average of 2 weeks
  Shoulder function will be measured by the disabilities of the arm, shoulder and hand (DASH) questionnaire, including the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). A higher score indicates greater disability.
Visual analogue scale (VAS) of shoulder pain and instability | Change from baseline visual analogue scale at the completion of 5-session intervention, an average of 2 weeks
  Shoulder pain and instability will be measured by visual analogue scale (VAS). Subjects need to mark the point that they feel represent their perception of their current state on a 10-cm line. Scores range from 0 (no symptom) to 100 (maximum symptom).

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No